CLINICAL TRIAL: NCT00707161
Title: A Prospective Phase II Study of Radiation Therapy and Concurrent Cisplatin Chemotherapy in the Treatment of Locally Advanced or Metastatic Malignant Melanoma
Brief Title: Radiation Therapy and Concurrent Cisplatin Chemotherapy for Locally Advanced or Metastatic Malignant Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: discontinued due to low enrollment
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI15461
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Cancer; Melanoma
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — Radiotherapy; Cisplatin; Drug Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All participants (Experimental)
  Interventions: Radiation: Radiation Therapy; Drug: Cisplatin; Procedure: Surgical resection

INTERVENTIONS:
Radiation: Radiation Therapy — Radiation therapy will be delivered concurrent with cisplatin chemotherapy as outlined in table 2. Radiation therapy dose will be 50 Gy (2.5 Gy per day, 5 days per week, for 20 treatments).
Drug: Cisplatin — Cisplatin dose will be 100 mg/m2 given i.v. every 3 weeks for a total of 2 doses (days 1 and 22) during radiation.
  Other Names: chemotherapy
Procedure: Surgical resection — Surgical resection of residual (or recurrent) melanoma for cure or for palliation may be performed following chemoradiation if deemed appropriate by the treating physicians (surgical resection may be planned following pre-operative chemoradiation or may be performed for salvage due to inadequate response to chemoradiation or for relapse following chemoradiation). Surgical resection will not be performed until at least 4 weeks following chemoradiation (unless deemed emergent by the treating physicians).
  Other Names: surgery

SUMMARY:
The study is a prospective phase II trial of radiation therapy concurrent with cisplatin chemotherapy in the treatment of locally advanced or metastatic melanoma in patients who are deemed to require radiation therapy by treating physicians for purposes of local control or palliation. Eligibility criteria include pathologically confirmed melanoma. Patients will undergo radiation therapy (20 treatments of 2.5 Gy for a total of 50 Gy) concurrent with cisplatin chemotherapy.

DETAILED DESCRIPTION:
This is a phase II, prospective trial designed to determine the response rate achieved with cisplatin delivered concurrent with radiation therapy in locally advanced or metastatic melanoma.

Radiation therapy will be delivered concurrent with cisplatin chemotherapy as outlined in table 2. Radiation therapy dose will be 50 Gy (2.5 Gy per day, 5 days per week, for 20 treatments). Cisplatin dose will be 100 mg/m2 given i.v. every 3 weeks for a total of 2 doses (days 1 and 22) during radiation.

Surgical resection of residual (or recurrent) melanoma for cure or for palliation may be performed following chemoradiation if deemed appropriate by the treating physicians (surgical resection may be planned following pre-operative chemoradiation or may be performed for salvage due to inadequate response to chemoradiation or for relapse following chemoradiation). Surgical resection will not be performed until at least 4 weeks following chemoradiation (unless deemed emergent by the treating physicians).

If the patient's tumor has inadequate response to chemoradiation then salvage therapies can be used as deemed appropriate by the treating physicians. In order to allow adequate response to radiation therapy, salvage therapies will not be utilized until at least 4 weeks following chemoradiation unless deemed emergent by the treating physicians.

ELIGIBILITY:
Inclusion criteria:

* Signed study-specific consent form prior to registration.
* Pathologically confirmed malignant melanoma.
* Measurable melanoma lesion deemed to require radiation by treating physicians for purposes of local control or palliation. The lesion may be the primary melanoma, a nodal metastasis, or a distant metastasis. Recurrent lesions are allowed.
* Lesion has to be measurable clinically or radiographically in 2 dimensions.
* Karnofsky Performance Scale (KPS) > 70.
* Laboratory values

  * White blood cells (WBC) > 3000/mm3
  * Absolute granulocyte count > 1,500
  * Platelets > 100,000/mm3
  * Total bilirubin < 2.0 x institutional upper limit of normal
  * AST or ALT (aminotransferase/alanine aminotransferase) < 2.5 x institutional upper limit of normal
  * Serum calcium < 1.3 x institutional upper limit of normal
  * Serum creatinine < 1.5 mg/dL or Creatinine clearance > 50 cc/min,calculated as follows: CCr = 0.85 x (140-age) x (weight in kg) 72 x serum creatinine in mg/dL

Exclusion criteria:

* Systemic therapy for malignant melanoma within one month preceding trial enrollment.
* Prior irradiation to the planned field.
* Concomitant chemotherapy (in addition to cisplatin) or biologic therapy is allowed.
* Significant infection or other co-existent medical condition which would prevent the use of full dose chemotherapy.
* Pre-existing sensory neuropathy (CTC 3.0 ≥ Grade II)
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Shrieve, MD, Principal Investigator — Huntsman Cancer Institute
Locations (2):
- United States (2):
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm (Radiation Therapy & Cisplatin): All patients will receive Radiation Therapy and Cisplatin for their melanoma. If appropriate patients will have surgical resection for residual or recurrent melanoma following chemoradiation.
Period: Overall Study
Arm/Group | Treatment Arm (Radiation Therapy & Cisplatin)
Started | 6 (3 deceased (1-Huntsman Cancer Institute, 2- LDS Hospital).)
Completed | 0
Not Completed | 6
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm (Radiation Therapy & Cisplatin): Radiation therapy given at 50 Gy, 20 fractions, for 4 weeks (2.5 Gy/day). Cisplatin given at 100mg/m2 i.v. every 3 weeks for a total of 2 doses (days 1 and 22) during radiation.
Arm/Group | Treatment Arm (Radiation Therapy & Cisplatin)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Melanoma Lesions
Description: Response rate of melanoma lesions was measured after treated with the trial agent.
Time Frame: 2005-2010
Population: Study terminated. Analysis not conducted.
Groups:
- Treatment Arm (Radiation & Cisplatin): Group of participants receiving Radiation and Cisplatin.
Arm/Group | Treatment Arm (Radiation & Cisplatin)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment Arm (Radiation Therapy & Cisplatin)
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Early termination due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes